CLINICAL TRIAL: NCT00346502
Title: Phase I/II Evaluation of Topical Application of 20% Betulinic Acid Ointment in the Treatment of Dysplastic Nevi With Moderate to Severe Dysplasia
Brief Title: Evaluation of 20% Betulinic Acid Ointment for Treatment of Dysplastic Nevi (Moderate to Severe Dysplasia)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tapas K. Das Gupta, PI, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0811
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Dysplastic Nevus Syndrome
MeSH Terms: conditions — Dysplastic Nevus Syndrome | interventions — Betulinic Acid

ARMS (1):
- Ointment (Experimental): Treatment will consist of four weeks of daily application of 20% BA ointment to the dysplastic nevi, after which it will be removed surgically and examined. A similar dysplastic nevi will be removed as a control. Four groups of patients will be enrolled. The first group will apply the ointment once a day, the second twice a day, the third three times a day, and the fourth four times a day.
  Interventions: Drug: 20% betulinic acid ointment; Drug: BA

INTERVENTIONS:
Drug: 20% betulinic acid ointment
Drug: BA — 20% Betulinic Acid Ointment
  Other Names: Betulinic Acid

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an experimental 20% betulinic acid ointment (BA ointment) as a treatment for dysplastic nevi with the potential to transform into melanoma.

DETAILED DESCRIPTION:
Approximately 200 patients may be enrolled and screened in order to find twenty-eight (28) patients who qualify to be involved in this research at UIC.

Dysplastic melanocytic nevus (DMN) is a histopathologic term implying a disordered proliferation of melanocytes associated with discontinuous and variable cellular atypia. DMN is graded into mild, moderate, and severe based on standard histological criteria. DMN is considered to be a likely precursor for melanoma, and individuals with DMN often have multiple instances of it scattered over their trunk and extremities. For this study, only DMN where the dysplasia is either moderate or severe will be included.

ELIGIBILITY:
Inclusion Criteria:

* All races are eligible for entry into the Study.
* All patients must have been histologically documented (by a punch biopsy) for dysplastic nevi with moderate to severe dysplasia (DMN). A similar biopsy proven DMN that will serve as the control needs to be available.
* Patients must be healthy and active in normal pursuits of life and be able to provide informed written consent.
* Localized dermatological conditions like psoriasis or actinic keratosis will not be an exclusion criteria.
* Patients must be ambulatory with an ECOG status < 2; they will not be hospitalized as part of the Study.
* All patients in this study will have, in addition to a normal clinical examination, a thorough skin examination. Whenever possible, periodic photographs of their lesions will be taken. Additional tests for all patients within 30 days of the initiation of topical application include urinalysis, a liver function test (LFT), and blood tests for complete blood count (CBC), BUN, and creatinine.

Exclusion Criteria:

* Women who are pregnant and/or nursing will be excluded. A pregnancy test will be performed on each pre-menopausal woman within two days of entry into the Study, and a negative pregnancy test must be recorded on the case report form prior to initiating use of the topical application.
* Patients who are being treated for other chronic debilitating diseases (cardiac, pulmonary, or any other organ specific diseases).
* Immuno-suppressed patients, either due to chemotherapy and radiation therapy or known immunodeficiency diseases (e.g., AIDS).
* Patients with other active malignancies within the past five years, excluding noninvasive skin or cervical carcinoma.
* Patients with any other serious medical or psychiatric illness that would prevent informed consent.
* Patients with extensive chronic skin diseases such as extensive psoriasis, atopic dermatitis, or xeroderma pigmentosa will be excluded from the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety | Weekly
  The development of any systemic toxicity (Grade 1 or greater) or Grade 3 local toxicity in 3 of 7 patients at any given dose level will result in the termination of all applications at that level; furthermore, no higher frequency of cohorts will be entered in the Study. This dose level is defined as a dose-limiting toxicity, with the maximum tolerated dose (MTD) being one dose level below.
Efficacy | 4-5 Weeks
  The response to the topical application of 20% betulinic acid ointment will be assessed histologically. Both the untreated control lesion and the betulinic acid treated lesion will be totally excised after four weeks (30 days) of treatment. Surgery to remove the lesions will take place between day 31 and day 37. The lesions will be processed for microscopic examination and will be examined by the Pathology Department of UIC/UIH. At the completion of the Study, all slides will be reviewed by a consultant dermato-pathologist.
  Evidence of regression, fibrosis, depigmentation, nuclear atypia, and apoptosis of melanocytes will be recorded for both untreated control and betulinic acid treated lesions. If the treated lesions demonstrate a significant difference in the points mentioned above, then the data will be quantitatively tabulated and interpreted.

CONTACTS AND LOCATIONS:
Overall Officials: Tapas K. Das Gupta, MD, PhD, DSc, Principal Investigator — University of Illinois at Chicago Medical Center
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States